CLINICAL TRIAL: NCT05701020
Title: Evaluation of Prevalence of Sexuality Alteration in Women With an Abnormal Pap Test
Acronym: EVASEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2019_843_0105
Record Dates: First submitted 2023-01-10; First posted 2023-01-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Sexual Dysfunction; Epidemiology
Keywords: Abnormal pap test; Sexual Dysfunction; Epidemiology
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult women with an abnormal pap test (Experimental)
  Interventions: Other: questionnary

INTERVENTIONS:
Other: questionnary — If agreeing to the protocol, ; patients will answered questions about sexual health during the gynecologic consultation

SUMMARY:
Human Papilloma virus is the most common sexual infection in women, which can leads to cervical lesion and cervical cancer. Pap test is recommanded in women of 25 years old until 65 years old in order to screen subclinic lesions and improve prognosis. Yet, scientific knowledge about chronic disease showed negative consequences on quality of life.

However, no study until now has striven to evaluate the consequences of an abnormal pap test on sexuality in adult women. The aim of this study is to evaluate if an abnormal pap test have an impact on the sexual functions in women because of the anxiety and psychological consequences of the diagnosis

ELIGIBILITY:
Inclusion Criteria:

* Adult women with an abnormal pap test.
* Diagnosis known 4 to 12 weeks before the appointment for colposcopy

Exclusion Criteria:

* Cervical cancer
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult women with an abnormal pap test
Enrollment: 90 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
% ofpositive response rate at the first question of the questionnaire | 18 months

SECONDARY OUTCOMES:
Number of causes of woman alteration sexual function alteration | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No